CLINICAL TRIAL: NCT05742555
Title: The Effect of Virtual Reality on Mental Well-Being and Quality of Life of Caregivers of Palliative Care Patients
Brief Title: Effect of Virtual Reality on Caregivers of Palliative Care Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Seda Karaman, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/451
Record Dates: First submitted 2023-02-03; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Mental Well-being; Quality of Life
Keywords: palliative care; caregiver; mental well-being; quality of life; virtual reality
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Other: Virtual reality intervention
- Control Group (No Intervention)

INTERVENTIONS:
Other: Virtual reality intervention — After the relatives of the patients included in the experimental group are informed about the study, they will be asked to fill in the Participant Information Form, Nottingham Health Profile (NSP) and Warwick-Edinburgh Mental Well-Being Scale (WEMIOÖ) after obtaining their permission. The virtual reality intervention will be applied to the caregivers at a suitable time of the day (when the patient's care and treatment is not intensive, the caregiver wishes). Different nature scenes (sea, forest, stream) with different types of music (classical music, nature sounds, relaxing music) will be watched for 10 minutes, 3 days a week. The application will be made for 4 weeks. At the end of this period, they will be asked to fill the NSP and WEMİOÖ again as a final test.
  Arms: Experimental Group

SUMMARY:
Due to advances in medical technology and accessible health services, the prognosis of diseases has improved and the need for care has increased, and primary caregivers have experienced the increased burden of caring for family members for a long time.

Because the patient is primarily responsible for continuing patient care in palliative care units and then at home, and especially because they have problems in psychological, social and financial support, caregivers within the family are considered as second-degree patients or occult patients.

Studies have shown that caregivers have a significant burden of care, therefore they experience serious depression, anxiety and physical problems, isolate themselves from society, and their quality of life decreases significantly.

In recent years, the use of virtual reality, which shows itself in different application areas in the field of health as a safe and useful system, has become widespread. Considering the use of virtual reality in the field of health; It is seen that it is mostly preferred for pain management, physical condition improvement, blood collection, burn treatment, and psychological disorder.

DETAILED DESCRIPTION:
Palliative care; It is a multidisciplinary approach that includes interventions to prevent complications and improve the quality of life of people with severe illness. Regardless of the level of development, palliative care units provide service in all countries.

The World Health Organization (WHO) stated that the aim of palliative care is not only to improve the quality of life of patients but also to support caregivers. Care burden is defined as negative subjective and objective consequences such as physical health problems, psychological distress, economic and social problems, deterioration of family relationships and loss of control.

The caregiver feels obliged to provide the patient's treatment, personal care and psychosocial support. The physical, economic and moral burden on the caregiver can negatively affect the caregiver socially, psychologically and physically over time.

Caregivers of palliative care patients have an important responsibility. The relationship between providing care and receiving care is in a delicate balance. caring for the patient; it turns into a dependent, intense, long-term and unilateral obligation. These adversely affect the caregiver's quality of life. In addition to the problems of patient care, caregivers also experience problems such as physical problems, fatigue, sleep disorders, behavioral changes, and loss of social roles. As a result, psychological and emotional disorders may occur in the caregiver. Eliminating the symptoms experienced by the caregiver and improving their quality of life are very important in the caregiving process.

The concept of virtual reality is defined as the combination of reality and imagination by transferring various realities to digital media and using special technological devices thanks to technological tools. The use of virtual reality in the field of health has become widespread and can be used for different purposes. Virtual reality application is most commonly used in patients for pain management, exercise training, burn treatments and psychological disorders. Looking at the literature, watching nature scenes; It has been observed that it reduces blood pressure and heart rate and respiratory rate in people, reduces stress and brain activity, and provides relaxation. No study has been found in the literature on caregivers who underwent virtual reality intervention. In this study, it is aimed to increase the mental well-being and quality of life of the relatives of patients who care for palliative care patients with virtual reality application.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Having the ability to read, understand and write Turkish,
* Does not have any psychiatric disorder and does not use drugs for it,
* Having a history of seizures,
* No migraine, vertigo, active nausea, vomiting, headache

Exclusion Criteria:

-Individuals with epilepsyIndividuals with vertigo

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-20 (Estimated); Primary Completion 2023-06-20 (Estimated); Study Completion 2023-08-20 (Estimated)

PRIMARY OUTCOMES:
Edinburgh Mental Well-Being Scale | through study completion, an average of 7 months
  Warwick-Edinburgh Mental Well-Being Scale (WEMIOÖ): WEMİOOS consists of 14 items and deals with the positive mental health of individuals, including psychological well-being and subjective well-being. A minimum of 14 points and a maximum of 70 points are taken from the scale. Higher scores mean higher psychological well-being. The scale is a 5-point Likert scale: "5: I totally agree, 4: I agree, 3: I somewhat agree, , 2: I don't agree, 1: I don't agree at all". All items of the scale are positive.
Nottingham Health Profile (NSP) | through study completion, an average of 7 months
  Nottingham Health Profile (NSP): It measures the health-related quality of life of individuals and the effect of their problems on social role functions. The first part of the scale with 38 items covers quality of life; The second part of 6 items measures the effects of problems on their functions in social roles. The first and second parts of the scale can be used independently of each other. In this study, the first part of the scale, consisting of 38 items and evaluating the quality of life answered as yes-no by the individual, will be used. It consists of 6 sub-dimensions: physical movement, sleep, pain, energy, emotional reactions and social isolation. The score of each sub-dimension ranges from 0-100. The total score is obtained by summing the scores of the 6 sub-dimensions. High scores indicate poor quality of life.